CLINICAL TRIAL: NCT03547635
Title: A Prospective, Multi-Center, Randomized, Parallel-group Study Comparing AMNIOEXCEL Plus Placental Allograft Membrane to a Marketed Comparator and Standard of Care Procedures in the Management of Diabetic Foot Ulcers
Brief Title: AMNIOEXCEL® Plus vs A Marketed Comparator vs SOC in the Management of Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T-AEPDFU-001
Record Dates: First submitted 2018-05-22; First posted 2018-06-06 (Actual); Results first posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This is a multicenter, randomized, parallel-group study comparing the outcomes associated with the use of AMNIOEXCEL Plus Placental Allograft Membrane, a marketed comparator and SOC alone in the management of diabetic foot ulcers (DFUs).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- AMNIOEXCEL Plus Amniotic Membrane (Experimental)
  Interventions: Other: AMNIOEXCEL Plus Amniotic Membrane
- A Marketed Comparator (Active Comparator)
  Interventions: Device: A Marketed Comparator
- Standard of Care (Other)
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: AMNIOEXCEL Plus Amniotic Membrane — AMNIOEXCEL Plus is a human placental-based tissue consisting of dehydrated, tri-layer Placental (Amnion/Chorion/Amnion) Allograft Membrane (T-PAM) layers. T-PAM is a minimally manipulated placental membrane product made from tissues donated by pre-screened mothers during planned C-sections and is intended for use as a wound covering. This product is an allograft tissue intended for homologous use for the repair, reconstruction and replacement of skin at the direction of a physician. AMNIOEXCEL Plus contains Human Cellular and Tissue Based Products (HCT/P) as defined by US FDA 21 CFR Part 1271. All donor recoveries are performed by BioDlogics, LLC, and adhere to the regulations regarding HCT/P recovery and the screening and testing of the tissue donor as verified through supplier audits.
  Arms: AMNIOEXCEL Plus Amniotic Membrane
Device: A Marketed Comparator — bi-layered skin substitute: the epidermal layer is formed by human keratinocytes and has a well-differentiated stratum corneum; the dermal layer is composed of human fibroblasts in a bovine Type I collagen lattice. It is indicated for use with standard therapeutic compression for the treatment of non-infected partial and full-thickness skin ulcers due to venous insufficiency of greater than 1-month duration and which have not adequately responded to conventional ulcer therapy. This product is also indicated for use with standard DFU care for the treatment of full-thickness neuropathic DFUs of greater than three weeks' duration which have not adequately responded to conventional ulcer therapy and which extend through the dermis but without tendon, muscle, capsule or bone exposure.
  Other Names: Apligraf®
  Arms: A Marketed Comparator
Other: Standard of Care — * Coban™
  * Conforming gauze
  * Optifoam® non-adhesive dressing
  * Cotton Gauze
  * Normal saline (liquid or gel)
  * Non-adhering dressings
  * Steristrips
  * An offloading boot (Pneumatic Short Leg Walker), as appropriate
  Arms: Standard of Care

SUMMARY:
This is a multicenter, randomized, parallel-group study comparing the outcomes associated with the use of AMNIOEXCEL Plus Placental Allograft Membrane, a marketed comparator and SOC alone in the management of diabetic foot ulcers (DFUs).

ELIGIBILITY:
Inclusion Criteria:

1. Have participated in the informed consent process and signed a study-specific informed consent document.
2. Be able and willing to comply with study procedures, including study visits, study dressing regimens, and compliance with study required offloading device.
3. Be ≥ 21 years of age.
4. Have Type I or Type II diabetes mellitus with Investigator-confirmed glycosylated hemoglobin (HbA1c) of ≤ 12%.
5. Have at least one diabetic foot ulcer Ulcer size (i.e., area) is > 1 cm2 and < 12 cm2.
6. Have adequate vascular perfusion of the affected limb

Exclusion Criteria:

1. The subject was previously randomized and treated under this clinical study protocol.
2. The study ulcer has features that necessitates surgical operating-room debridement and/or penetrates to capsule/tendon/bone.
3. The subject is unable to safely ambulate with the use of a study required offloading boot.
4. The subject has suspected or confirmed gangrene or wound infection of the study ulcer.
5. The subject has suspected or confirmed osteomyelitis.
6. In the opinion of the Investigator, the subject has received or is scheduled to receive during study participation, a medication or treatment which is known to interfere with or affect the rate and quality of wound healing
7. The subject has a history of bone cancer or metastatic disease of the affected limb, radiation therapy to the foot, or has had chemotherapy prior to signing the Informed Consent Form for trial participation.
8. The subject is currently pregnant or is actively trying to conceive.
9. In the opinion of the Investigator, the subject is unable to comply with the treatment regimen
10. In the opinion of the Investigator, the subject has a history of, or is currently diagnosed with, any illness or condition, other than diabetes, that could interfere with wound healing.
11. In the opinion of the Investigator, the subject has a condition that could inhibit wound healing.
12. The subject has ulcers secondary to a disease other than diabetes.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2019-02-26 (Actual); Study Completion 2019-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Knowlton, MS CRA, Study Director — Integra LifeSciences Corporation
Locations (7):
- United States (7):
  - California 1, Fresno, California
  - California 3, Fresno, California
  - California 2, Los Angeles, California
  - Georgia 1, Gainesville, Georgia
  - Illinois 1, Springfield, Illinois
  - New Jersey 1, Toms River, New Jersey
  - Texas 1, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Snyder RJ, Shimozaki K, Tallis A, Kerzner M, Reyzelman A, Lintzeris D, Bell D, Rutan RL, Rosenblum B. A Prospective, Randomized, Multicenter, Controlled Evaluation of the Use of Dehydrated Amniotic Membrane Allograft Compared to Standard of Care for the Closure of Chronic Diabetic Foot Ulcer. Wounds. 2016 Mar;28(3):70-7. PMID 26978860
- [Background] Martinson M, Martinson N. A comparative analysis of skin substitutes used in the management of diabetic foot ulcers. J Wound Care. 2016 Oct 1;25(Sup10):S8-S17. doi: 10.12968/jowc.2016.25.Sup10.S8. PMID 27681811
- [Background] Snyder RJ, Cardinal M, Dauphinee DM, Stavosky J. A post-hoc analysis of reduction in diabetic foot ulcer size at 4 weeks as a predictor of healing by 12 weeks. Ostomy Wound Manage. 2010 Mar 1;56(3):44-50. PMID 20368673

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care: Standard of Care: • Coban™
  * Conforming gauze
  * Optifoam® non-adhesive dressing
  * Cotton Gauze
  * Normal saline (liquid or gel)
  * Non-adhering dressings
  * Steristrips
  * An offloading boot (Pneumatic Short Leg Walker), as appropriate
Period: Overall Study
Arm/Group | AMNIOEXCEL Plus Amniotic Membrane | A Marketed Comparator | Standard of Care
Started | 41 | 38 | 37
Completed | 33 | 31 | 29
Not Completed | 8 | 7 | 8
Not completed — Adverse Event | 5 | 2 | 3
Not completed — Lost to Follow-up | 1 | 3 | 4
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Withdrawal By PI | 0 | 1 | 0
Not completed — Withdrawal by Sponsor | 0 | 0 | 1
Not completed — Errant Randomization before Treatment | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (All Randomized Subjects)
Groups:
- Total: Total of all reporting groups
Arm/Group | AMNIOEXCEL Plus Amniotic Membrane | A Marketed Comparator | Standard of Care | Total
Number analyzed (Participants) | 41 | 38 | 37 | 116
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (11.32) | 60.5 (11.10) | 59.6 (11.03) | 59.1 (11.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 6 | 35
  Male | 25 | 25 | 31 | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 18 | 20 | 52
  Not Hispanic or Latino | 27 | 20 | 17 | 64
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 1 | 1 | 6
  White | 37 | 37 | 36 | 110
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 41 | 38 | 37 | 116

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Meeting Criteria of Complete Wound Closure, as Assessed by the Investigator at or Before Week 12 of the Treatment Phase, Which is Confirmed Closed Two Weeks Later.
Description: Complete wound closure is defined as complete skin re-epithelialization that is without drainage or dressing requirements.
Time Frame: Wound closure assessed up to week 12 and confirmed 2 weeks later; only participants with wound closure at or before Week 12 and who maintained closure in follow-up reported
Measure: Count of Participants; unit: Participants
Arm/Group | AMNIOEXCEL Plus Amniotic Membrane | A Marketed Comparator | Standard of Care
Number analyzed (Participants) | 41 | 38 | 37
Participants | 12 | 16 | 8

ADVERSE EVENTS:
Time Frame: Date of randomization through last treatment visit which could be on or before 12 weeks of treatment.
Description: Note: A subject in the Marketed Comparator group was randomized, but not treated. This subject was removed from the study by the investigator is not counted in the AE/SAE group.
Arm/Group | AMNIOEXCEL Plus Amniotic Membrane | A Marketed Comparator | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/37 | 0/37
Serious Adverse Events (participants affected / at risk) | 2/41 | 1/37 | 2/37
Other Adverse Events (participants affected / at risk) | 4/41 | 5/37 | 9/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AMNIOEXCEL Plus Amniotic Membrane (N=41) | A Marketed Comparator (N=37) | Standard of Care (N=37)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic Foot Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AMNIOEXCEL Plus Amniotic Membrane (N=41) | A Marketed Comparator (N=37) | Standard of Care (N=37)
Cellulitis (Infections and infestations) | 2 (2) | 2 (2) | 3 (3)
Diabetic Foot Infection (Infections and infestations) | 2 (2) | 3 (3) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators are barred from publishing or disclosing results until a multicenter publication is published or until a period of 24 months after study completion passes, whichever comes first.

DOCUMENTS (2):
  • Study Protocol (2018-11-05): https://cdn.clinicaltrials.gov/large-docs/35/NCT03547635/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/35/NCT03547635/SAP_001.pdf